CLINICAL TRIAL: NCT00482378
Title: An Open-Label, Pilot Study of Samarium - Sm 153 Lexidronam (Quadramet) in Patients With Relapsed or Refractory Multiple Myeloma and Bone Pain
Brief Title: Samarium Sm 153 Lexidronam Pentasodium Combined With Zoledronic Acid or Pamidronate in Treating Patients With Relapsed or Refractory Multiple Myeloma and Bone Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546769; P30CA015083 (NIH); MC048B (Other: Mayo Clinic Cancer Center); 261-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm; Pain
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; pain
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Pain | interventions — Pamidronate; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sm 153 lexidronam (Experimental)
  Interventions: Drug: Pamidronate; Drug: Zoledronic acid; Radiation: Sm 153 lexidronam

INTERVENTIONS:
Drug: Pamidronate — 90 mg by IV monthly.
  Other Names: Aredia
Drug: Zoledronic acid — 4 mg by IV monthly.
  Other Names: Zometa
Radiation: Sm 153 lexidronam — 0.5 mCi/kg or 1 mCi/kg by IV.
  Other Names: Sm 153 lexidronam consists of radioactive samarium and a tetraphosphonate chelator, ethylenediaminetetramethylenephosphonic acid (EDTMP).

SUMMARY:
RATIONALE: Radioactive drugs, such as samarium Sm 153 lexidronam pentasodium, may carry radiation directly to cancer cells and not harm normal cells. Zoledronic acid and pamidronate may help relieve bone pain caused by multiple myeloma. Giving samarium Sm 153 lexidronam pentasodium together with zoledronic acid or pamidronate may be an effective treatment for multiple myeloma.

PURPOSE: This phase I/II trial is studying the side effects and best dose of samarium Sm 153 lexidronam pentasodium when given together with zoledronic acid or pamidronate and to see how well it works in treating patients with relapsed or refractory multiple myeloma and bone pain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of samarium Sm 153 lexidronam pentasodium in combination with zoledronic acid or pamidronate disodium in patients with relapsed or refractory multiple myeloma and bone pain. (Phase I)
* Determine the clinical response in patients treated with these regimens. (Phase II)

Secondary

* Determine the effect of these regimens on changes in patient-reported bone pain levels.

OUTLINE: This is a multicenter, open-label, pilot, phase I, dose-escalation study of samarium Sm 153 lexidronam pentasodium followed by a phase II study.

* Phase I: Patients receive samarium Sm 153 lexidronam pentasodium IV over 1 minute on day 1. Patients also receive zoledronic acid IV over 15 minutes or pamidronate disodium IV over 2-4 hours on day 1 and then monthly thereafter in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of samarium Sm 153 lexidronam pentasodium until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive samarium Sm 153 lexidronam pentasodium at the MTD determined in phase I and zoledronic acid or pamidronate disodium as in phase I.

Bone pain is assessed periodically.

After completion of study treatment, patients are followed every 3-6 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Relapsed or refractory disease, meeting 1 of the following criteria:

    * Recurrent disease after stem cell transplantation
    * Recurrent or progressive disease despite treatment with ≥ 1 standard regimen (e.g., an alkylating agent plus glucocorticoid and/or the combination of vincristine, doxorubicin hydrochloride, and dexamethasone)
* Measurable or evaluable disease, defined by at least 1 of the following:

  * Monoclonal protein ≥ 1.0 g by serum protein electrophoresis
  * Monoclonal protein ≥ 200 mg by 24-hour urine electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)
* Patients must have already undergone hematopoietic stem cell collection, if believed to be a transplant candidate OR not eligible for a hematopoietic stem cell transplant

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 (ECOG PS 3 allowed if secondary to pain)
* ANC ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8.0 g/dL (transfusions allowed)
* Creatinine ≤ 3 mg/dL
* Calcium < 15 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after completion of study therapy
* No impending long bone fracture
* No active malignancy except for nonmelanoma skin cancer or carcinoma in situ of the cervix or breast
* No uncontrolled infection
* No other co-morbidity that would interfere with the patient's ability to participate in this trial
* No known hypersensitivity to any of the components of samarium Sm 153 lexidronam pentasodium or bisphosphonates

PRIOR CONCURRENT THERAPY:

* Recovered from all prior surgery, radiotherapy, or other antineoplastic therapy
* More than 4 weeks since prior melphalan or other myelosuppressive agents
* More than 2 weeks since prior nonmyelosuppressive agents (e.g., thalidomide or high-dose corticosteroids)
* More than 30 days since prior and no other concurrent investigational therapy
* No prior samarium Sm 153 lexidronam pentasodium or strontium chloride Sr 89
* No concurrent external beam radiotherapy
* No concurrent high-dose corticosteroids

  * Concurrent chronic steroids (maximum dose of 20 mg/day prednisone equivalent) allowed for disorders other than myeloma (i.e., adrenal insufficiency or rheumatoid arthritis)
  * Low-dose steroids allowed for replacement or inhalation therapy
* No other concurrent medications, including any of the following:

  * Cytotoxic chemotherapy
  * Systemic antineoplastic therapy including, but not limited to, immunotherapy, hormonal therapy, or monoclonal antibody therapy
  * Prophylactic hematopoietic growth factors

    * Hematopoietic growth factors allowed for established cytopenia therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2005-03-21 (Actual); Primary Completion 2007-05-22 (Actual); Study Completion 2008-12-02 (Actual)

PRIMARY OUTCOMES:
Toxicity (Phase I) | 12 weeks
Confirmed clinical response of serum and urine monoclonal protein (Phase II) | 12 weeks

SECONDARY OUTCOMES:
Response (Phase I) | 12 weeks
Bone pain response (Phase II) | 12 weeks
Toxicity (Phase II) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States